CLINICAL TRIAL: NCT02952053
Title: Can Myotonometry Quantify Dry Needling Effectiveness on Myofascial Trigger Points?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other); Universidad San Jorge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 134b
Record Dates: First submitted 2016-10-29; First posted 2016-11-02 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2016-10

CONDITIONS: Muscle Tone Abnormalities
Keywords: Myofascial Trigger Points; Dry needling; Myotonometry

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling into MTrPs. (Experimental): MTrP Group: Deep Dry Needing into the medial Myofascial Trigger Point of the soleus muscle.
  Interventions: Device: MTrP Group
- Dry Needling within Taut Band (Active Comparator): TB Group: Deep Dry Needling distal to Myofascial Trigger Point of the soleus muscle (in the same taut band; out of MTrPs).
  Interventions: Device: TB Group

INTERVENTIONS:
Device: MTrP Group — Deep Dry Needling into the site of the latent medial Myofascial Trigger Point of the soleus muscle.
  1 session in soleus muscle. 10 fast in and fast out needle insertions.
  Arms: Dry Needling into MTrPs.
Device: TB Group — Deep Dry Needling distal to Myofascial Trigger Point but into the same taut band.
  1 session in soleus muscle. 10 fast in and fast out needle insertions.
  Arms: Dry Needling within Taut Band

SUMMARY:
The main objective of this study is to assess effects of Dry Needling into Myofascial Trigger Point compared Dry Needling into Taut Band point based on the outcomes of myotnometric measurement in healthy subjects.

Hypothesis: Deep Dry Needling of the latent medial Myofascial Trigger Point (MTrP) of the soleus muscle will achieve changes in myotonometric measures compared to Deep Dry Needling of the Taut Band of the soleus muscle.

DETAILED DESCRIPTION:
Methods:

It is a double-blinded randomized clinical trial where subjects are healthy volunteers from the city of Toledo older than 18 years.

There will be a MTrP Group (dry needling into the medial MTrP of soleus muscle) and a TB Group (dry needling distal to the MTrP but into the taut muscle band of soleus muscle). The intervention will be a unique session.

Intervention:

Dry needling technique will be performed by locating the taut band and the Myofascial Trigger Point. Depending on the group, a thin needle (0,32x40mm) is introduced 10 times (fast in and fast out) directly within the Myofascial Trigger Point or within the Taut Band.

Assessment:

Myoton device is a simple and portable tool to obtain quantitative and objective assessments of mechanical properties of muscle tone. Myoton has been adopted to characterize the viscoelastic properties of skeletal muscle as tissue displacement when a mechanical perturbation is applied to the muscle.

The device incorporates a probe and an acceleration sensor. The probe was kept perpendicular with its end touching the muscle belly. 10 mechanical impacts (with a duration of 15 ms, a force of 0.4 N and a local deformation in the order of a few millimetres) are delivered to MTrP and TB points.

Outcome measures:

Outcome measures will include myotonometric measurements (frecuency, stiffness and decrement) and they will be evaluated before, at 10 min and 1 week after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-40 years.
* Healthy volunteers.
* Presence of a latent medial MTrP of the soleus muscle.
* Being able to provide written informed consent.
* Being able to follow instructions and realize clinical tests.

Exclusion Criteria:

* Any history of ipsilateral lower limb severe injury or intervention (e.g. fracture, surgical intervention).
* Pain or musculoskeletal injury, ligament injury, tendonitis or plantar fasciitis in the ipsilateral leg for six months previous to the intervention.
* Peripheral or central nervous system neurological disease.
* Altered sensitivity in the treatment area.
* Treatment of a myofascial trigger point in the sural triceps in the six months previous to the intervention.
* Changes in physical activity which would have affected muscle tone during the study.
* Fear of needles.
* No tolerance to pain caused by dry needling.
* No continuance commitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-12-12 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Oscillation Frequency. | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  This outcome measure is obtained by a device named MyotonPro. The frequency of the damped oscillations characterizes the muscle tone.
Change in Stiffness. | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  This outcome measure is obtained by a device named MyotonPro. Stiffness reflects the resistance of the muscle to the force deforming the muscle.
Change in Decrement (elasticity). | Pre-intervention (Day 1); After intervention (Day 1); Follow up (1 week after intervention).
  This outcome measure is obtained by a device named MyotonPro.The logarithmic decrement of the damping oscillations characterizes muscle elasticity which is the ability of the muscle to restore its initial shape after contraction.

SECONDARY OUTCOMES:
Pain perception after intervention using Visual Analogical Scale. | After intervention (Day 1).
  Pain perception after intervention using Visual Analogical Scale (VAS).
Number of Local Twitch Responses. | During intervention (Day 1).
  Number of local twitch responses during intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Gomez Soriano, PhD, Study Director — University of Castilla-La Mancha; María Ortiz Lucas, PhD, Study Director — Universidad San Jorge; Carolina Jiménez Sánchez, MSc, Principal Investigator — Universidad San Jorge
Locations (1):
- Universidad San Jorge, Villanueva de Gállego, Spain

IPD SHARING:
Plan to Share IPD: No